CLINICAL TRIAL: NCT01702155
Title: A Phase I/II Study of DFP 10917 Given by Continuous Infusion in Patients With Relapsed or Refractory Acute Leukemia
Brief Title: Phase I/II Study of DFP-10917 in Patients With Acute Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Delta-Fly Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D11-11002
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — DFP-10917

ARMS (1):
- DFP-10917 (Experimental): 1. 7-day continuous infusion (in the vein): Starting dose 4 mg/m^2
  2. 14-day continuous infusion (in the vein): Starting dose 10 mg/m^2
  3. Phase II Only: 6 mg/m^2 for the 14-day continuous infusion (in the vein)
  Interventions: Drug: DFP-10917

INTERVENTIONS:
Drug: DFP-10917

SUMMARY:
The purpose of this study is to determine the safety and efficacy of DFP-10917 given via continuous 7 or 14 day infusion to patients with acute leukemias (AML or ALL).

DETAILED DESCRIPTION:
This study will determine the safety and efficacy of DFP-10917 in patients with AML or ALL. The Phase I dose-escalation portion of the study will determine the highest tolerable dose and regimen (7 or 14 day continuous infusion) based on safety data in patients with refractory or relapsed AML or ALL. The phase II portion will investigate the safety and efficacy of DFP-10917, at the dose and regimen to be determined in the Phase I portion, in patients with refractory or relapsed AML.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically-confirmed acute leukemia, refractory or relapsed after standard therapy for the disease or for which conventional systemic chemotherapy is not reliably effective or no effective therapy is available Phase II Only: Patient must have histologically or pathologically confirmed diagnosis of AML based on WHO classification that is refractory after standard therapy, or for which conventional systemic chemotherapy is not reliably effective, or no effective therapy is available. Patients aged 60 years or older with newly diagnosed AML who are not eligible for, or who refuse, standard care are also eligible.
2. Aged ≥ 18 years.
3. ECOG Performance Status of 0, 1 or 2.
4. Adequate clinical laboratory values (i.e., plasma creatinine <= 1.5 x upper limit of normal (ULN) for the institution, bilirubin <=1.5 x ULN, alanine transaminase (ALT) and aspartate transaminase (AST) <= 2.5 x ULN).
5. Absence of CNS involvement by leukemia.
6. Absence of uncontrolled intercurrent illnesses, including uncontrolled infections, cardiac conditions, or other organ dysfunctions.
7. Signed informed consent prior to the start of any study specific procedures.
8. Women of child-bearing potential must have a negative serum or urine pregnancy test. Male and female patients must agree to use acceptable contraceptive methods for the duration of the study and for at least one month after the last drug administration.

Exclusion Criteria:

1. The interval from prior treatment to time of study drug administration is < 2 weeks for cytotoxic agents or < 5 half-lives for noncytotoxic agents. Exceptions: Use of hydroxyurea is allowed before the start of study and may be administered up to day 5 of the first cycle.
2. Any >grade 1 persistent clinically significant toxicities from prior chemotherapy.
3. Extensive prior radiotherapy to more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation.
4. Any concomitant condition that in the opinion of the investigator could compromise the objectives of this study and the patient's compliance.
5. A pregnant or lactating woman.
6. Current malignancies of another type. Exceptions: Patients may participate if they have previously treated and currently controlled prostate cancer, adequately treated in situ cervical cancer and basal cell skin cancer or other malignancies with no evidence of disease for 2 years or more.
7. Patient has acute promyelocytic leukemia (APL).
8. Patients with known HIV, HBV or HCV infection (note: testing for these infections is not required).
9. Documented or known clinically significant bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Kantarjian HM, Jabbour EJ, Garcia-Manero G, Kadia TM, DiNardo CD, Daver NG, Borthakur G, Jain N, Waukau JB, Kwari MI, Ravandi F, Anderson BD, Iizuka K, Jin C, Zhang C, Plunkett WK. Phase 1/2 study of DFP-10917 administered by continuous intravenous infusion in patients with recurrent or refractory acute myeloid leukemia. Cancer. 2019 May 15;125(10):1665-1673. doi: 10.1002/cncr.31923. Epub 2019 Jan 22. PMID 30668890
- See also: Publication of Study Results — https://www.ncbi.nlm.nih.gov/pubmed/30668890